CLINICAL TRIAL: NCT03041272
Title: Aggressive Incidents in Medical Settings Study
Acronym: AIMS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1609018379
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nurses and nursing personnel: All registered nurses and assistive nursing personnel, including patient care associates (PCAs) , patient care technicians (PCTs), clinical technicians (CTs), primary employment on the study unit, minimum of 24 hours per week of employment on study unit.

SUMMARY:
The purpose of this study is to identify the incidence rate and characteristics of aggressive behavior perpetrated by patients and visitors in inpatient medical units and to understand the role of missed care events, professional quality of life and self-efficacy in relationship to aggressive events.

DETAILED DESCRIPTION:
This prospective cohort study will examine the incidence of and outcomes associated with patient and visitor aggressive behavior towards nursing staff practicing on medical inpatient units. Staff on each unit will be informed about the AIMS study and all eligible nursing staff will be invited to participate in the study. After completing the informed consent nursing staff will be asked to complete the baseline demographic form and survey on professional quality of life. For the data collection phase of the study consented participants will be educated on use of the AIM log and provided with scenarios to practice AIM log use. Consented staff will carry event counters and use the AIM log for all shifts worked over the next 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All registered nurses and assistive nursing personnel, including patient care associates (PCAs) , patient care technicians (PCTs), clinical technicians (CTs),
* primary employment on the study unit,
* minimum of 24 hours per week of employment on study unit.

Exclusion Criteria:

* Any registered nurse or assistive nursing personnel working less than 24 hours per week,
* whose primary employment is on a unit not involved in the study or float-pool / centralized resource staff who do not have a primary employment unit,
* any nursing staff member still on orientation or working with an orientee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study of nursing staff on inpatient medical units will seek to enroll all RN's and nursing assistive personnel meeting eligibility criteria from three units at Yale New Haven hospital.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
unit-level incidence rate of patient and visitor physical aggression | 2 weeks
  Event counters and logs will be used to record aggressive event data and will be recorded on the AIM log over the 2 week data collection period. The midnight census on each unit will be recorded over the 2 week data collection period and the average number of occupied beds will be used in the calculation of this rate. The formula used will be:
  (Number of physical aggression events recorded in 2 week period) divided by (Average number of occupied beds in 2 week period)
unit-level incidence rate of patient and visitor verbal aggression | 2 weeks
  Event counters and logs will be used to record aggressive event data and will be recorded on the AIM log over the 2 week data collection period. The midnight census on each unit will be recorded over the 2 week data collection period and the average number of occupied beds will be used in the calculation of this rate. The formula used will be:
  (Number of verbal aggression events recorded in 2 week period) divided by (Average number of occupied beds in 2 week period)

SECONDARY OUTCOMES:
To describe the characteristics of patient and visitor events involving aggressive behavior toward nursing staff in inpatient medical settings. | 2 weeks
  Data on aggressive events and patient characteristics will be aggregated from the AIM Logs, Descriptive statistics will be used to summarize events including: frequency of each type of event (verbal, physical or both); severity of event; perpetrator of event; precipitant of event; target of event, objects or body parts used, interventions and consequences of events. In addition written descriptions of events will be qualitatively summarized.
risk of missed care events | 2 weeks
  Missed care event data will be retrieved from aggressive incident and management logs (AIM log). Analysis will include the standard descriptive statistics. An evaluation of the risk of missed care events will be carried out using initially a dichotomous identification of a missed care event (defined as any reason for missed care) using chi-square tests to identify significant differences by characteristics of aggressive events. Categories of missed care involving direct physical intervention (ambulation, turning, mouth care, feeding, bathing/skin care); psychosocial intervention (patient teaching, emotional support); medication related interventions (assessing effectiveness, within 5 minutes of prn medication); or assessment or monitoring (vital signs, Intake & Output documentation, blood glucose monitoring) will be used in analyses to describe missed care types.
Professional Quality of Life Scale | 2 weeks
  The relationship of aggressive event exposure rates to scores on the Professional Quality of Life Scale (ProQOL) will be analyzed using chi-square tests to identify significant differences between stratified groups and logistic regression will be used to evaluate differences between high vs low exposure groups (high defined as greater than the median level of exposure in subjects) and professional quality of life scores with adjustment for potential confounders (age, gender, role, length of experience, length of work on unit).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Iennaco, Principal Investigator — Yale School of Nursing
Locations (3):
- United States (3):
  - Middlesex Hospital, Middletown, Connecticut
  - Yale New Haven Hospital- St. Raphael, New Haven, Connecticut
  - Yale New Haven Hospital Primary Care Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No